CLINICAL TRIAL: NCT04809324
Title: Intra-operative Gross Examination Versus Frozen Section for Achievement of Adequate Margin in Patients Undergoing Surgery for Oral Cavity Squamous Cell Carcinoma: A Randomized Controlled Trial
Brief Title: Gross Examinations Versus Frozen Section for Assessment of Surgical Margins in Oral Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr.Pankaj Chaturvedi (Other)
Responsible Party: Sponsor-Investigator, Dr.Pankaj Chaturvedi, Dr Pankaj Chaturvedi ,Prof. and Surgeon, Dept of Head Neck Surgery, Tata Memorial Centre
Organization: Tata Memorial Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: protocol no 3541; CTRI/2021/03/032015 (Registry Identifier: Clinical Trials registry of India)
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Oral Cavity Cancer
Keywords: Oral squamous Cell carcinoma; frozen section; local recurrence
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Frozen Sections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: patient and the treating clinician will not be aware of the randomisation allocation(gross examination or frozen section) prior to resection of the tumour specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gross examination (Experimental): measurement of the surgical margins will be done by the surgeon in the operating room using sterile scale after resection of the primary tumor .
  Interventions: Procedure: Gross examination of the resection specimen
- Frozen section (Active Comparator): frozen section examination of surgical margins will be done by the pathologist.
  Interventions: Procedure: Frozen section

INTERVENTIONS:
Procedure: Gross examination of the resection specimen — measurement of the surgical margin by the operating surgeon using sterile scale, margins <7mm will be revised on table
  Arms: Gross examination
Procedure: Frozen section — frozen section evaluation of the specimen by the pathologist
  Arms: Frozen section

SUMMARY:
Surgical margin is a significant prognostic factor in oral cavity squamous cell carcinoma (OCSCC)[1,2,3]. Intra-operative frozen section (FS) has been routinely used by the surgeons to achieve adequate surgical margins. However published literature has failed to show a conclusive benefit of FS in improving oncological outcomes(4-7). The overall identification rate of the inadequate margins by FS is variable with figures in the literature ranging from25-34%.(8-10)

Revision of margins based on FS is widely practiced in centers where facility for FS is available. However this has not shown to significantly improve local control when compared to cases in which FS was not utilized , in a comparative study done at Tata memorial Hospital(TMH) (5) More-over FS is a costly procedure, and sparsely available in resource- poor countries. In a recently conducted retrospective study of 1237 patients conducted at TMH, the cost benefit ratio of FS for assessment of margin is as low as 12:1(11). In another prospective study performed at the same center , investigators found that gross examination (GE) of margins by the surgeons was as effective as FS, and achievement of gross 7mm margin all around the tumor obviated the need for FS (12). In a recent meta-analysis of 8 studies that looked at the utility of frozen section and had uniformity in frozen section analysis and definition of close margins, they concluded that revision of margins based on FS does not improve oncological outcomes and further prospective studies are needed to explore this contentious issue (13). With this background, a prospective RCT is planned to explore if gross examination by surgeon and subsequent revision of margin (if necessary) is an equally effective alternative to Frozen section based revision in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven treatment naïve cases of OCSCC who are planned for curative surgery with en-bloc removal of the tumor with adequate margin
2. In detail assessment of the primary tumor is possible pre-operatively
3. Written informed consent
4. Age more than 18 years

Exclusion Criteria:

1. Multifocal disease
2. Clinically evident field cancerization
3. Previous treatment for oral cavity cancer - Surgery /chemo or radiotherapy -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1206 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
local recurrence free survival (LRFS) between two arms | 2 years
  To determine the difference between the local recurrence free survival (LRFS) between intra operative gross examination by the surgeon compared with microscopic examination using frozen sections by the pathologist for the assessment of surgical margin in patients undergoing surgery for OCSCC.
  Local recurrence will be defined as - tumor recurrence at the same subsite or or at margins of previous surgery &/ reconstruction with or without nodal recurrence /distant metastases withing two years after completion of the treatment.
  - Isolated regional &/or distant metastasis without recurrence at local site will be recorded however it will not be considered as the event for measuring LRFS

SECONDARY OUTCOMES:
Accuracy of gross examination | 5 years
  To determine the accuracy of intra operative gross examination by the surgeon compared with microscopic examination of frozen sections by the pathologist for the assessment of surgical margin as compared to the final histopathology report as the gold standard.
Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of GE and FS for the assessment of surgical margin | 5years

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Chaturvedi, MS, Principal Investigator — Tata Memorial Centre
Locations (3):
- India (3):
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - ACTREC,Advanced Centre for Treatment, Research and Education in Cancer, Navi Mumbai, Raigad
  - Mahamana Pandit Madan Mohan Malaviya Cancer Centre, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal To achieve aims in the approved proposal for individual participant data meta-analysis.
  Proposals should be directed to chaturvedi.pankaj@gmail.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Looser KG, Shah JP, Strong EW. The significance of "positive" margins in surgically resected epidermoid carcinomas. Head Neck Surg. 1978 Nov-Dec;1(2):107-11. doi: 10.1002/hed.2890010203. PMID 755803
- [Background] Loree TR, Strong EW. Significance of positive margins in oral cavity squamous carcinoma. Am J Surg. 1990 Oct;160(4):410-4. doi: 10.1016/s0002-9610(05)80555-0. PMID 2221245
- [Background] Chen TY, Emrich LJ, Driscoll DL. The clinical significance of pathological findings in surgically resected margins of the primary tumor in head and neck carcinoma. Int J Radiat Oncol Biol Phys. 1987 Jun;13(6):833-7. doi: 10.1016/0360-3016(87)90095-2. PMID 3583852
- [Background] Pathak KA, Nason RW, Penner C, Viallet NR, Sutherland D, Kerr PD. Impact of use of frozen section assessment of operative margins on survival in oral cancer. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Feb;107(2):235-9. doi: 10.1016/j.tripleo.2008.09.028. Epub 2008 Dec 13. PMID 19071037
- [Background] Mair M, Nair D, Nair S, Dutta S, Garg A, Malik A, Mishra A, Shetty Ks R, Chaturvedi P. Intraoperative gross examination vs frozen section for achievement of adequate margin in oral cancer surgery. Oral Surg Oral Med Oral Pathol Oral Radiol. 2017 May;123(5):544-549. doi: 10.1016/j.oooo.2016.11.018. Epub 2016 Dec 7. PMID 28159583
- [Background] Kovacs AF. Relevance of positive margins in case of adjuvant therapy of oral cancer. Int J Oral Maxillofac Surg. 2004 Jul;33(5):447-53. doi: 10.1016/j.ijom.2003.10.015. PMID 15183407
- [Background] Scholl P, Byers RM, Batsakis JG, Wolf P, Santini H. Microscopic cut-through of cancer in the surgical treatment of squamous carcinoma of the tongue. Prognostic and therapeutic implications. Am J Surg. 1986 Oct;152(4):354-60. doi: 10.1016/0002-9610(86)90304-1. PMID 3766863
- [Background] DiNardo LJ, Lin J, Karageorge LS, Powers CN. Accuracy, utility, and cost of frozen section margins in head and neck cancer surgery. Laryngoscope. 2000 Oct;110(10 Pt 1):1773-6. doi: 10.1097/00005537-200010000-00039. PMID 11037842
- [Background] Ord RA, Aisner S. Accuracy of frozen sections in assessing margins in oral cancer resection. J Oral Maxillofac Surg. 1997 Jul;55(7):663-9; discussion 669-71. doi: 10.1016/s0278-2391(97)90570-x. PMID 9216496
- [Background] Ribeiro NF, Godden DR, Wilson GE, Butterworth DM, Woodwards RT. Do frozen sections help achieve adequate surgical margins in the resection of oral carcinoma? Int J Oral Maxillofac Surg. 2003 Apr;32(2):152-8. doi: 10.1054/ijom.2002.0262. PMID 12729775
- [Background] Datta S, Mishra A, Chaturvedi P, Bal M, Nair D, More Y, Ingole P, Sawakare S, Agarwal JP, Kane SV, Joshi P, Nair S, D'Cruz A. Frozen section is not cost beneficial for the assessment of margins in oral cancer. Indian J Cancer. 2019 Jan-Mar;56(1):19-23. doi: 10.4103/ijc.IJC_41_18. PMID 30950438
- [Background] Chaturvedi P, Datta S, Nair S, Nair D, Pawar P, Vaishampayan S, Patil A, Kane S. Gross examination by the surgeon as an alternative to frozen section for assessment of adequacy of surgical margin in head and neck squamous cell carcinoma. Head Neck. 2014 Apr;36(4):557-63. doi: 10.1002/hed.23313. Epub 2013 Jun 14. PMID 23765548
- [Background] Bulbul MG, Tarabichi O, Sethi RK, Parikh AS, Varvares MA. Does Clearance of Positive Margins Improve Local Control in Oral Cavity Cancer? A Meta-analysis. Otolaryngol Head Neck Surg. 2019 Aug;161(2):235-244. doi: 10.1177/0194599819839006. Epub 2019 Mar 26. PMID 30912991